CLINICAL TRIAL: NCT02584621
Title: Web-Supported Adolescent Motivational Enhancement to Reduce Alcohol Use
Brief Title: Web-Based Adolescent Motivational Enhancement Study
Acronym: Web-AME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seattle Children's Hospital (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Carolyn McCarty, Principal Investigator, Seattle Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 3679948; 1R21AA023050-01A1 (NIH)
Record Dates: First submitted 2015-10-21; First posted 2015-10-22 (Estimated); Last update posted 2017-10-05 (Actual); Status verified 2017-10

CONDITIONS: Alcohol Risk Behaviors; Health Care Services Quality of Care

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Check Yourself App With Feedback (Experimental): Participants complete Check Yourself, an electronic health screening app and receive personalized, motivational feedback on their health behaviors prior to their visit with their health provider. Key components of Check Yourself include the provision of age normative feedback, goal setting strategies, and strategies to highlight discrepancies. Health providers receive a summary report of health risk behaviors from Check Yourself prior to the visit.
  Interventions: Behavioral: Check Yourself App with Feedback
- Usual Care (No Intervention): Participants are asked to complete health risk screening questions on a tablet computer. No personalized feedback is provided to adolescents and primary care providers do not receive a summary report of the adolescent's health risk behaviors.

INTERVENTIONS:
Behavioral: Check Yourself App with Feedback
  Arms: Check Yourself App With Feedback

SUMMARY:
The proposed study is a randomized controlled trial that compares the effectiveness of an electronic personalized health screening app incorporating motivational feedback (i.e. "Check Yourself") to usual care among moderate to high risk alcohol users. The purpose of this study is to determine whether Check Yourself is more effective than usual care in reducing alcohol consumption and binge drinking and improving quality of care among adolescents receiving school-based health clinic services.

ELIGIBILITY:
Inclusion Criteria:

* Eligible individuals will be 13-18 years old who are able to read and comprehend English.
* Participants who indicate alcohol use consistent with moderate to high risk on the Check Yourself App.

Exclusion Criteria:

Individuals will be excluded from the study if:

* They do not meet age requirements
* Do not have a study visit at a participating school-based health clinic
* Lack the means to complete follow-up interviews (i.e. have neither telephone or internet access)
* Are not able to read or comprehend English

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 148 (Actual)
Dates: Start 2015-11; Primary Completion 2017-02 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Alcohol Use Frequency and Quantity | 2 months
  Adolescent reported level for alcohol risk behaviors at 2 months adjusting for baseline level. Specific alcohol behaviors include: 1) number of days in which alcohol was consumed in the past 30 days; 2) number of alcoholic drinks typically consumed per occasion; and 4) maximum number of alcoholic drinks consumed during one drinking episode.
Adolescent report of whether alcohol was counseled on during health provider visit | 1 day

SECONDARY OUTCOMES:
Marijuana Use Frequency and Quantity | 2 months
  Adolescent reported level for marijuana risk behaviors at 2 months adjusting for baseline level. Specific marijuana behaviors include: 1) number of days in which marijuana was used in the past 30 days; and 2) number of hours high on a typical day of marijuana use.
Adolescent Satisfaction with Care | 1 day
  Adolescent satisfaction with care will be assessed using the total score on the 8-item Client Satisfaction Questionnaire (CSQ-8) at 1-day follow-up.
Interval Receipt of Care for Substance Use | 2 months
  Dichotomous variable indicating receipt of any follow-up care to address substance use identified at baseline.
Adolescent Substance Use Problem Recognition | 1 day & 2 months
  Adolescent reported recognition of alcohol and/or marijuana use as a problem (5-point scale).
Motivation for Substance Use Behavior Change | 1 day & 2 months
  Adolescent reported motivation to change alcohol use and/or marijuana use using a readiness to change scale (4-point scale).

OTHER OUTCOMES:
Number of non-substance use health risk behaviors | 2 months
  Total count of non-substance use health risk behaviors at 2-month follow-up (score range=0-11) adjusted by total number of baseline health risk behaviors which include (with risk cut-off): during a typical day >2 sugar-sweetened beverages consumed or <3 servings of fruits/vegetables consumed; during a typical week <3 days with 60+ minutes of exercise; during a typical school day >3 hours of screen time; during a typical night <7 hours of sleep; not "always" using seatbelt; not "always" using helmet when bicycling; having driven/ridden in a car with a driver under the influence of substances; not using birth control during last sexual intercourse; not "always" using a condom; and a score of >10 on the Patient Health Questionnaire (PHQ-9).
Adolescent perceived support from their health care provider | 1 day
  The total score on the Health Care Climate Questionnaire (HCCQ) will be used to assess adolescent self-report of perceived autonomy support from their health care provider.
Adolescent report of whether marijuana/other drug use was counseled on during health provider visit | 1 day

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Interagency Teen Health Center, Seattle, Washington
  - Garfield Teen Health Center, Seattle, Washington
  - Nathan Hale Teen Health Center, Seattle, Washington